CLINICAL TRIAL: NCT07110480
Title: Combination of Equisetum Arvense and Pea for the Management of Chronic Pain
Brief Title: Combination of Equisetum Arvense and Palmitoylethanolamide (PEA) for the Management of Patients With Chronic Pain in a Before-after Study
Acronym: Assonal®️PEA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: noiVita Srls (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 704/CE; noivita srls (Other: noivita srls)
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Chronic Pain (Back / Neck); Pain (Visceral, Somatic, or Neuropathic); Pain Management
MeSH Terms: conditions — Chronic Pain; Pain; Agnosia | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AssonalPEA (Experimental): The product evaluated in the following protocol is a new formulation containing 600 mg of PEA and 300 mg of Equisetum arvense L. (Assonal®️PEA) per tablet to reduce the symptoms of chronic pain. Enrolled patients will be advised to take 1 or 2 tablets per day at any time of the day, preferably swallowed with a sip of water. The product should be stored in a cool, dry place, away from localized heat sources and sunlight, and protected from moisture. It is advisable to keep the tablets in the blister pack until ready to take them.
  Interventions: Dietary Supplement: Supplement

INTERVENTIONS:
Dietary Supplement: Supplement — The enrolled patient was advised to take 1 to 2 tablets daily at any time, preferably with a sip of water, as directed by the pharmaceutical company. In detail, starting with the distribution of Assonal®️PEA (T0) by the principal investigator, patients took 2 tablets per day (1 in the morning and 1 in the evening) for the first 15 days of treatment (T1). Treatment continued with 1 tablet per day until the end of the clinical study (T3).

SUMMARY:
Chronic pain is a type of pain that lasts or recurs for a period of more than three months. Due to the physical, psychological, and socio-relational consequences of chronic pain for the person experiencing it, it has been recognized as a true pathology in itself. In fact, it interferes with daily activities, causing depression, mistrust, and a general sense of malaise. Acetaminophen or nonsteroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen or naproxen, are generally used as the first line of treatment for chronic pain. NSAIDs are able to reduce inflammation, which is often linked to the pathology and exacerbates it, as well as alleviate chronic pain. However, if taken in high doses or over a prolonged period, NSAIDs can cause serious side effects, such as irritation of the gastrointestinal mucosa, an increased tendency to bleed, kidney problems, and a high risk of cardiovascular abnormalities. In this context, the present study aims to identify a new treatment useful for managing chronic pain. For this purpose, patients suffering from chronic pain, attending the Alessandria Hospital Company, aged between 18 and 80, and using acetaminophen in the previous 3 months, would be enrolled. Enrolled patients would be administered oral tablets containing 600 mg of palmitoylethanolamide (PEA) and 300 mg of Equisetum arvense L. In detail, recent research has highlighted the anti-inflammatory and immunomodulatory role of PEA, which has a neuroprotective effect, acting on several molecular targets in the central and peripheral nervous systems . Furthermore, PEA is an endogenous agonist of the endocannabinoid system, acting on CB1 and CB2 receptors, allowing proper nerve transmission and regulating the sensation of chronic pain . In addition, numerous studies have described the biological effects of Equisetum A.L. extract, as it plays an important role in the oxidative stress response mechanism and in the activation of SIRT1, which mediates chronic pain Based on this evidence, in the present study, PEA and Equisetum A.L. are administered simultaneously to evaluate their synergistic effect on the modulation of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 80 years of age.
* Pain beyond 3 months, even intermittent, timing is necessary to have a pattern of chronic pain.
* Signature of informed consent.
* Paracetamol use in the last 3 months.

Exclusion Criteria:

* Drug treatment for chronic pain (e.g., acetyl-L-carnitine, tricyclic antidepressants, opioids, antiepileptics) would lead to incorrect interpretation of data.
* Pharmacological treatment for arthritis pain would lead to an incorrect interpretation of the data.
* Psychiatric disorders or cognitive dysfunction in patients with these disorders could result in the completion of questionnaires that are not useful for the final assessment.
* Concomitant severe brain damage.
* Tumours or terminal illnesses.
* Pregnancy or lactation.
* Alcohol or substance abuse.
* Allergies or intolerance to the product as it would cause serious adverse side effects

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | - T0: baseline - T1: after 14 days - T2: after 30 days - T3: after 60 days
  The primary endpoint was the reduction of perceived pain, which was measured using the NPRS at T0, T1, T2, T3. The NPRS (or NRS scale) is a one-dimensional 11-point scale that assesses the intensity of pain in adults, including chronic pain conditions due to rheumatic diseases]. The scale is composed of a horizontal line, with an interval ranging from 0 to 10, corresponding to "no pain" and "worst imaginable pain", respectively. The NPRS scale can be easily administered both verbally (for example, also by telephone) and graphically.
Verbal Rating Scale | - T0: baseline - T1: after 14 days - T2: after 30 days - T3: after 60 days
  The Verbal Rating Scale (VRS) is a pain scale consisting of a list of descriptors that identify the degree of pain intensity. Generally, the scale ranges from "no pain" to "severe pain" or "very intense pain," passing through a series of intermediate adjectives that should gradually capture the nuances of intensity of the painful experience, such as "mild," "moderate," and "severe."

SECONDARY OUTCOMES:
measurement of patient perception versus drug treatment | - T0: baseline - T1: after 14 days - T2: after 30 days - T3: after 60 days
  The measurement of patient perception versus drug treatment, which will be measured with the GPE, a scale that assesses patient perception using a 7-point Likert scale. This is a subjective assessment in which the patient indicates how much they feel improved or worsened compared to before treatment (1: Very much worse; 2: Moderately worsened; 3: Slightly improved; 4: No change; 5: Slightly improved; 6: Moderately improved; 7: Much improved). This scale is widely used in clinical trials and clinical practice to assess the effectiveness of therapeutic interventions, particularly in musculoskeletal and rehabilitation settings.
quantification and description of perceived pain | - T0: baseline - T1: after 14 days - T2: after 30 days - T3: after 60 days
  The quantification and description of perceived pain will be assessed using the SF-MPQ. It is a self-assessment questionnaire that al-lows you to have an accurate description of the quality and intensity of the pain that the subject is experiencing. There are 78 items di-vided into 20 subgroups that refer to 4 main categories: the sensory class, the affective class, the valuative class and the miscellaneous class. The SF-MPQ also includes the Pain Intensity Index (PPI) of the standard MPQ and a visual analogue scale (VAS).
Measuring quality of life | - T0: baseline - T1: after 14 days - T2: after 30 days - T3: after 60 days
  Measuring quality of life, described with the EURO-QoL-5D-5L or EQ-5D-5L. The instrument consists of: a 5-dimensional descriptive system (mobility, self-care ability, habitual activities, pain/discomfort, and anxiety/depression), each of which involves a three-point rating scale (no problem=1 point; some problem=2 points; persistent problem=3 points); and a VAS that requires the subject to answer the question, "How healthy do you feel today?" A score of 0 corresponds to the worst health status ever, while 100 equals the best perceived health level. It is possible to combine the scores of the two sections and determine an overall score

CONTACTS AND LOCATIONS:
Locations (1):
- DAIRI, Alessandria, AL, Italy

IPD SHARING:
Plan to Share IPD: No